CLINICAL TRIAL: NCT03601923
Title: Phase 2 Proof-of-Concept Trial Testing the PARP Inhibitor Niraparib in Patients With Pancreatic Cancer Harboring Deficiencies in Homologous Recombination DNA Repair
Brief Title: Niraparib in Patients With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Principal Investigator, James Cleary, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-207
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): * Niraparib will be administered orally once daily
  * Palliative radiation therapy to a small field >1 week prior to Day 1 of study treatment
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib belongs to a class of anti-cancer agents known as PARP (poly ADP ribose polymerase) inhibitors. PARP is a protein in the body that repairs damage to DNA (one of the building blocks of a cell). In cells that are rapidly growing, such as cancer cells, blocking repair of DNA may be of benefit, since it will cause the cell to die.
  Niraparib will be given at an initial dose of 200mg or 300 mg by mouth once daily depending on the patient's platelet count and weight at the start of the trial.
  Other Names: Zejula

SUMMARY:
This research study is studying an investigational therapy as a possible treatment for pancreatic cancer.

The drugs involved in this study are:

-Niraparib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease.

The FDA (the U.S. Food and Drug Administration) has not approved niraparib for this specific disease but it has been approved for other uses.

Niraparib belongs to a class of anti-cancer agents known as PARP (poly ADP ribose polymerase) inhibitors. PARP is a protein in the body that repairs damage to DNA (one of the building blocks of a cell). In cells that are rapidly growing, such as cancer cells, blocking repair of DNA may be of benefit, since it will cause the cell to die.

In this research study, the investigators are looking to test the effectiveness of niraparib in patients with pancreatic cancer. The trial is focused on pancreatic cancer patients that have marker, a mutation in a DNA repair gene, suggesting that their cancer might be susceptible to niraparib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed advanced pancreatic adenocarcinoma that is not curable with standard approaches. Patients with metastatic pancreatic cancer and unresectable pancreatic cancer are eligible.
* Patients must have molecular characteristics that fulfill one of the following requirements:

  * Germline deleterious BRCA1, BRCA2, PALB2, CHEK2 or ATM mutations. Germline variants of unknown significance are not eligible.
  * Somatic mutation in BRCA1, BRCA2, PALB2, CHEK2 or ATM
  * Germline and somatic testing need to be performed in CLIA approved laboratories. Deleterious genetic mutations should either be described in the literature or felt by expert opinion (in consultation with the principal investigator) to interfere with the protein's DNA repair function. The somatic mutational testing can be performed on tissue samples taken from any time in the patient's pancreatic cancer history.
* Patients must have received at least one line of treatment for their cancer prior to enrolling on the trial.
* Patients who had investigator assessed progression on an oxaliplatin-containing regimen (such as FOLFOX or FOLFIRINOX) are not eligible for the trial.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Age ≥ 18 years. As no dosing or adverse event data are currently available in participants < 18 years of age, children are excluded from this study.
* ECOG performance status of 0 or 1 (see Appendix A)
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 9g/dL
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 × institutional ULN -OR-
  * Creatinine clearance ≥ 30 mL/min/1.73 m2 for participants with serum creatinine levels above the institutional ULN
  * Albumin ≥ 2.7 g/dL
* Female participants must have a negative serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  --≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range (>35μlU/mL) upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See Section 5.5 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. --Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
* Male participant agrees to use an adequate method of contraception (see Section 5.5 for a list of acceptable birth control methods) starting with the first dose of study treatment through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Ability to swallow and retain oral medication.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must be willing to undergo a pre-treatment fresh tumor biopsy. The biopsy requirement can be waived only after discussion with the principal investigator.
* Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.

Exclusion Criteria:

* Participants who have had cytotoxic chemotherapy, radiotherapy, immunotherapy, biologic therapy, or other investigational therapy within 2 weeks prior to entering the study or those who have not recovered to ≤ CTCAE (version 5.0) Grade 1 or baseline from adverse events due to agents administered more than 2 weeks earlier (with the exceptions of alopecia and peripheral neuropathy).
* Participants must not have received investigational therapy administered ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior initiating protocol therapy.
* Participants who have received oral targeted therapy or tyrosine kinase inhibitor (TKI) therapy within 5 half-lives or 2 weeks of study entry, whichever is shorter.
* Participants who have been previously treated with a PARP inhibitor.
* Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
* Participants who have undergone major surgery ≤ 3 weeks prior to initiating protocol therapy. Participants must have sufficiently recovered from adverse events caused by the procedure as judged by the treating investigator.
* Participants with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with a history of brain metastases that have been treated, are no longer taking corticosteroids, and have been stable on imaging for ≥ 4 weeks following the last date of treatment are permitted.
* History of hypersensitivity to compounds of similar chemical or biologic composition to niraparib or its excipients.
* Participants must not be immunocompromised. Participants with prior splenectomy are allowed.
* Participants must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Participants must not have current evidence of any condition, therapy, or laboratory abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study or interfere with the participant's participation for the full duration of the study treatment or that makes it not in the best interest of the participant to participate.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV-positive participants are ineligible because these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Participants with a clinically significant gastrointestinal disorder that in the opinion of the treating investigator could impact the absorption of the study drug, including but not limited to malabsorption syndrome or major resection of the stomach or bowels.
* Participants with a history of a clinically relevant second primary malignancy within the past 2 years. Exceptions include: resected basal and squamous cell carcinomas of the skin and completely resected carcinoma in situ of any type.
* Participants must not be on anticoagulant therapy unless the treating investigator has deemed it safe to temporarily hold to facilitate the collection of the pre-treatment tumor biopsy.
* Participant must not have received colony stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 month
  Progression-free survival is defined as the time from registration to documented disease progression or death from any cause, whichever occurs first. Subjects who have not experienced an event of interest by the time of analysis will be censored at the date of the last disease assessment without progression.

SECONDARY OUTCOMES:
Overall response rate will be measured by RECIST criteria. | 2 years
Overall Survival Rate | 2 years
  Overall survival is defined as the time from registration to death from any cause, and subjects who are thought to be alive at the time of final analysis will be censored at the last date of contact.
Evaluation of the safety and tolerability of niraparib as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Cleary, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No